CLINICAL TRIAL: NCT03914898
Title: Effect of Nurse-Led Intervention Programme on Compassion Fatigue, Burnout, Compassion
Brief Title: Effect of Nurse-Led Intervention Programme Professional Quality of Life and Psychological Distress in Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Neslihan Partlak Günüşen, Associate professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3109-GOA
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Compassion Fatigue
Keywords: burnout; compassion fatigue; nursing; psychological distress
MeSH Terms: conditions — Compassion Fatigue; Burnout, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse led intervention group (Experimental): The program was four sessions; It took about 1.5-2 hours. The intervention group was divided into two groups. The author who administered the intervention previously led nurse support groups, is also an active educator in psychiatry and mental health nursing, and has training in cognitive behavioral therapy.
  The group sessions were based on cognitive restructuring techniques.
  Interventions: Other: Nurse led intervention group
- Control Group (No Intervention): No intervention was applied to the control group during the study.

INTERVENTIONS:
Other: Nurse led intervention group — This program is based on cognitive restructuring tecniques.
  Arms: Nurse led intervention group

SUMMARY:
Nurses are at risk in terms of burnout and empathic fatigue. Therefore, efforts to protect the mental health of nurses are very important. It is stated that the studies conducted are mostly descriptive and not interventional.

In addition, the evidence levels of interventional studies are low.

DETAILED DESCRIPTION:
Aim:The aim of this study is to reduce nurses' psychological distress, burnout and secondary trauma stress.

Design This single-blind randomized controlled trial design was used. Measurements were made before, after and 6 months after Participants and Settings The study was perform at a hospital in Turkey. Intervention program was applied in 4 week. 84 nurses meeting the criteria were invited to the program.48 nurses agreed to participate. Nurses were randomly assigned groups.

Sample Size the sample was calculated with the open epi program. The sample size was calculated as 20 per group.

Intervention The program was created to reduce nurses' psychological distress, and improve the professional quality of life.

The intervention programme were four sessions. The Intervention group was divided into two groups. Intervention were applied in a comfortable room in the hospital. Interventions were based on cognitive behavioral approach.

Outcome measures The outcomes were compassion fatigue, burnout and compassion satisfaction, psychological distress.

These variables were evaluated by the Professional Quality of Life Scale (ProQOL-IV). The GHQ-12 is a scale surveying psychological distress observed within the last few weeks.

Data collection Research data were collected before, immediately after, and six months after intervention.

Validity and reliability Measuring tools showing good psychometric properties were used to ensure validity and reliability. Volunteer participants were randomly assigned to groups, and the intention-to-treat approach was used for data analysis. The study has been reported in accordance with the CONSORT 2010 Statement principles.

Ethical considerations Permission was obtained from the relevant university, and written permission was obtained from the hospital. The participants were informed, all participants gave written consent.

Data analysis Mann Whitney U test, and Friedman analysis was used. All analyses were made on an intention-to-treat approach. Missing data were compensated for using the last observation method carried forward.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who responded to the questionnaires received a score on compassion fatigue higher than the mean score (20 points)
* Nurses who worked at clinics and had at least six months of experience

Exclusion Criteria:

* Nurses who responded to the questionnaires received a score on compassion fatigue lower than the mean score (20 points)
* head nurses

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline compassion fatigue at 1 and 6 months assessed by compassion fatigue subscale of Professional quality of life scale | Data collected before the program starts and one months after the end of the program and six months
  The compassion fatigue subscale of ProQOL-IV includes 10-items. Completion of the compassion fatigue subscale involves selecting response choices on a 0 (never) to 5 (very often) likert scale. 0-50 points can be taken from the compassion fatigue subscale. There is no cut-point. A number of items required reverse coding so that high scores on all items indicate high compassion fatigue.
Change from baseline burnout at 1 and 6 months assessed by burnout subscale of Professional quality of life scale | Data collected before the program starts (pretest) and one months after the end of the program and six months
  The burnout subscale of ProQOL-IV includes 10-items. Completion of the burnout subscale involves selecting response choices on a 0 (never) to 5 (very often) likert scale. 0-50 points can be taken from the burnout subscale. There is no cut-point. A number of items required reverse coding so that high scores on all items indicate high burnout.
Change from baseline compassion satisfaction at 1 and 6 months assessed by compassion satisfaction subscale of Professional quality of life scale | Data collected before the program starts (pretest) and one months after the end of the program and six months
  The compassion satisfaction subscale of ProQOL-IV includes 10-items. Completion of the compassion satisfaction subscale involves selecting response choices on a 0 (never) to 5 (very often) likert scale. 0-50 points can be taken from the compassion satisfaction subscale. There is no cut-point. A number of items required reverse coding so that high scores on all items indicate high compassion satisfaction.

SECONDARY OUTCOMES:
Change from baseline psychological distress at 1 and 6 months assessed by general health questionnaire | Data collected before the program starts (pretest) and one months after the end of the program and six months
  The GHQ-12 is a scale surveying psychiatric symptoms observed within the last few weeks. The items were evaluated on a 4-point likert-type scale. Scoring was as follows (a) and (b), 0 points; (c) and (d), 1 point; and the total possible score ranged between 0 and 12 points. The General Health Questionnaire-12 (GHQ-12) states that the nurses who score 2 and above risky.

CONTACTS AND LOCATIONS:
Locations (1):
- Neslihan Günüşen, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marine A, Ruotsalainen J, Serra C, Verbeek J. Preventing occupational stress in healthcare workers. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD002892. doi: 10.1002/14651858.CD002892.pub2. PMID 17054155
- [Background] Potter P, Deshields T, Berger JA, Clarke M, Olsen S, Chen L. Evaluation of a compassion fatigue resiliency program for oncology nurses. Oncol Nurs Forum. 2013 Mar;40(2):180-7. doi: 10.1188/13.ONF.180-187. PMID 23448743
- [Background] Pfaff KA, Freeman-Gibb L, Patrick LJ, DiBiase R, Moretti O. Reducing the "cost of caring" in cancer care: Evaluation of a pilot interprofessional compassion fatigue resiliency programme. J Interprof Care. 2017 Jul;31(4):512-519. doi: 10.1080/13561820.2017.1309364. Epub 2017 May 4. PMID 28471255
- [Background] Yilmaz G, Ustun B, Gunusen NP. Effect of a nurse-led intervention programme on professional quality of life and post-traumatic growth in oncology nurses. Int J Nurs Pract. 2018 Dec;24(6):e12687. doi: 10.1111/ijn.12687. Epub 2018 Aug 5. PMID 30079550
- [Background] Gunusen NP, Ustun B. An RCT of coping and support groups to reduce burnout among nurses. Int Nurs Rev. 2010 Dec;57(4):485-92. doi: 10.1111/j.1466-7657.2010.00808.x. Epub 2010 Sep 7. PMID 21050201
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860